CLINICAL TRIAL: NCT01706107
Title: Canadian Multicenter Observational Study of Tysabri in Early Relapsing Remitting Multiple Sclerosis Patients
Brief Title: Canadian Multicenter Observational Study of Tysabri in Early Relapsing Remitting Multiple Sclerosis Participants
Acronym: COSTAN
Status: Terminated | Type: Observational
Why Stopped: Due to on-going enrollment challenges
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-TYS-12-10333
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the study is to evaluate the impact of early treatment with Tysabri in Relapsing Remitting Multiple Sclerosis (RRMS) participants on their quality of life (QoL) as measured by Multiple Sclerosis Impact Scale-29 (MSIS-29) over 2 years. The secondary objectives of the study are: to evaluate the impact of early treatment with Tysabri in RRMS participants over 2 years on the following: annualized relapse rate (ARR), Expanded Disability Status Scale (EDSS), work productivity, quality of life (QoL) by EuroQol 5-Dimension questionnaire (EQ-5D), QoL by Subject Global Assessment of Wellbeing visual analog scale (VAS) and to evaluate clinical disease-free status (relapses, EDSS) over 2 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent.
* Documented diagnosis of Relapsing Multiple Sclerosis (McDonald 2010 Criteria).
* Must have an Expanded Disability Status Scale (EDSS) score from 0 to 4.0, inclusive.
* Must satisfy the approved therapeutic indications for Tysabri as per Product Monograph.
* Must either be treatment naïve or have been treated with disease modifying therapy DMT(s) (such as, but not limited to, Avonex, Betaseron, Rebif, Copaxone, Extavia, Tecfidera and/or Gilenya) for ≤5 years total prior to date of informed consent.
* Decision to treat with Tysabri must precede enrollment.

Key Exclusion Criteria:

* Any prior treatment with Tysabri.
* Contraindications to treatment with Tysabri as described in the Product Monograph.
* History of progressive multifocal leukoencephalopathy (PML) or other opportunistic infections, or an increased risk for such infections.
* History of diagnosis of Primary Progressive Multiple Sclerosis [PPMS] and/or Secondary Progressive Multiple Sclerosis [SPMS].
* Receiving immunomodulatory or immunosuppressive therapy.
* Prior history of immunosuppressive use (mitoxantrone, azathioprine, methotrexate, cyclophosphamide, mycophenolate, cladribine, rituximab).
* Immunocompromised at the time of enrollment.
* Known active malignancies (subjects with cutaneous basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* Women breastfeeding, pregnant, or planning to become pregnant; women who are not post-menopausal or surgically sterile who are unwilling to practice contraception.
* Inability to comply with study requirements.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who choose to participate in the study will receive a thorough description of the study protocol and an informed consent document describing the study and the risks and benefits of participating. Recruitment will continue until approximately 150 patients have been enrolled in the study at approximately 15 sites across Canada.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2015-10-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Multiple Sclerosis Impact Scale-29 (MSIS-29) | Baseline, Months 12 and 24
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.

SECONDARY OUTCOMES:
Change from Baseline in Annualized Relapse Rate | Baseline, Months 12 and 24
  A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement.
Change from Baseline in Expanded Disability Status Scale (EDSS) | Baseline, Months 12 and 24
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Change from Baseline in Work Productivity and Activity Impairment | Baseline, Months 12 and 24
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Change from Baseline in EuroQol 5-Dimension (EQ-5D) | Baseline, Months 12 and 24
  The EQ-5D is a self-administered questionnaire consisting of 5 sets of 3 questions pertaining to specific health states (i.e., mobility, self-care, pain, usual activities, anxiety), and a visual analog scale that records the respondent's self-rated health from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in Patient Global Assessment of Wellbeing Visual Analog Scale | Baseline, Months 12 and 24
  Patient Global Assessment of Wellbeing measures quality of life on a 100 mm Visual Analog Scale (VAS) where 0 is the worst imaginable health state and 100 is the best imaginable health state.
Percentage of participants with Clinical Disease-Free Status | Baseline, Months 12 and 24
  Freedom from clinical disease activity is defined as the percentage of participants with no relapse and no EDSS progression, defined as a 1-point change from baseline. EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- Canada (11):
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dalhousie MS Research Unit, Halifax, Nova Scotia
  - Cape Breton Regional Hospital, Sydney, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique Neuro-Outaouais, Gatineau, Quebec
  - Neuro Rive-Sud, Greenfield Park, Quebec
  - CHUM - Hopital Notre Dame, Montreal, Quebec
  - McGill University - MNI, Montreal, Quebec
  - CHUS - Hopital Fleurimont, Sherbrooke, Quebec